CLINICAL TRIAL: NCT03552549
Title: A Randomized Phase II/III Trial of SCH 54031 PEG12000 Interferon Alfa-2b (PEG Intron) vs. INTRON®A as Adjuvant Therapy for Melanoma
Brief Title: SCH 54031 PEG12000 Interferon Alfa-2b (PEG Intron, MK-4031) vs. INTRON®A (SCH 30500, MK-2958) as Adjuvant Therapy for Melanoma (C98-135, MK-4031-002)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This study was closed to enrollment prematurely due to sub-optimal accrual.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C98135; MK-4031-002 (Other: Merck Protocol Number); C98-135 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2b; Introns; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-Intron (Experimental): Participants with stage III node positive cutaneous melanoma will receive subcutaneous PEG-Intron (6.0 ug/kg weekly) for 2 years post-surgery.
  Interventions: Biological: PEG-Intron
- INTRON A (Experimental): Participants with stage III node positive cutaneous melanoma will receive intravenous INTRON A (20 million international units [MIU]/m^2/day, 5 days a week) for 4 weeks followed by subcutaneous INTRON A (10 MIU/m^2 three times per week) for 48 weeks post-surgery.
  Interventions: Biological: INTRON A

INTERVENTIONS:
Biological: PEG-Intron — Polyethylene glycol (PEG)12000 Interferon alfa 2-b subcutaneous injection.
  Other Names: peginterferon alfa-2b, SCH 54031, MK-4031
  Arms: PEG-Intron
Biological: INTRON A — Interferon alfa-2b, recombinant for intravenous injection.
  Other Names: interferon alfa-2b, SCH 30500, MK-2958
  Arms: INTRON A

SUMMARY:
This is a Phase II/III randomized, controlled, multicenter, open-label study designed to assess the safety, efficacy, and impact on quality of life of PEG Intron (MK-4031) and INTRON® A (MK-2958) and the pharmacokinetics of PEG Intron when given as adjuvant (after surgery) therapy in participants with resected (surgically removed) Stage III node-positive cutaneous melanoma.

DETAILED DESCRIPTION:
This study was closed to enrollment prematurely due to sub-optimal accrual. Participants who were enrolled prior to enrollment closure were allowed to continue to receive study drug; these participants were followed for safety only.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically documented primary cutaneous melanoma meeting one of the following staging criteria:

  * Primary melanoma of any stage in the presence of N1 regional lymph node metastases detected at elective lymph node dissection or sentinel node biopsy, with clinically inapparent regional lymph node metastasis (any pTN1M0).
  * Clinically apparent N1 or N2a regional lymph node involvement synchronous with primary melanoma of T1-4 (any pTN1-2aM0).
  * Regional lymph node recurrence at any interval after appropriate surgery for primary melanoma of any depth (any primary tumor [pT], r N1-2a M0).
* Participants must have had all known disease completely resected with adequate surgical margins within 56 days prior to randomization into the study
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants must have adequate hepatic, renal and bone marrow function as defined by the following parameters obtained within 14 days prior to initiation of study treatment:

  * Hematology: white blood cells (WBC) ≥3,000 cells/µL and hemoglobin ≥9 g/dL.
  * Renal and hepatic function: serum creatinine <2.0 mg/dL; aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) <2 times upper limit of laboratory normal (ULN); and serum bilirubin <2 times ULN
* Participants must sign and date a voluntary informed consent form before study entry, be willing to participate in this study and agree to complete all follow-up assessments.

Exclusion Criteria:

* Participants who have received any prior chemotherapy, immunotherapy hormonal or radiation therapy for melanoma.
* Participants who have evidence of distant or non-regional lymph node metastases, in-transit metastases, or positive lymph nodes with an unknown primary.
* Participants whose disease cannot be completely surgically resected because of gross extracapsular extension.
* Participants who have previously received interferon for any reason.
* Participants who have severe cardiovascular disease, i.e., arrhythmias requiring chronic treatment, congestive heart failure (New York Heart Association [NYHA] Class III or IV) or symptomatic ischemic heart disease.
* Participants who have a history of neuropsychiatric disorder requiring hospitalization.
* Participants with thyroid dysfunction not responsive to therapy.
* Participants with uncontrolled diabetes mellitus.
* Participants with a history of prior malignancy within the past 5 years other than surgically cured non-melanoma skin cancer or cervical carcinoma in situ.
* Participants who have a history of seropositivity for human immunodeficiency virus (HIV).
* Participants who are pregnant, lactating, or of reproductive potential and not practicing an effective means of contraception.
* Participants with active and/or uncontrolled infection, including active hepatitis.
* Participants with a medical condition requiring chronic systemic corticosteroids.
* Participants who are known to be actively abusing alcohol or drugs.
* Participants who have received any experimental therapy within 30 days prior to randomization in this study.
* Participants who have not recovered from the effects of recent surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 1998-08-05 (Actual); Primary Completion 2001-02-19 (Actual); Study Completion 2001-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG-Intron: Participants with stage III node positive cutaneous melanoma received subcutaneous PEG-Intron (6.0 ug/kg weekly) for up to 24 months post-surgery
- INTRON A: Participants with stage III node positive cutaneous melanoma received intravenous INTRON A (20 million international units [MIU]/m^2/day, 5 days a week) for 4 weeks followed by subcutaneous INTRON A (10 MIU/m^2 three times per week) for up to 12 months post-surgery
Period: Overall Study
Arm/Group | PEG-Intron | INTRON A
Started | 63 | 63
Treated | 62 | 62
Completed | 10 | 11
Not Completed | 53 | 52
Not completed — Disease progression | 25 | 17
Not completed — Adverse event in first 12 months | 12 | 8
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Unknown (no reason provided) | 4 | 2
Not completed — Not in participant's best interest | 2 | 1
Not completed — Did not complete study treatment | 2 | 3
Not completed — Did not meet eligibility criteria | 1 | 0
Not completed — Administrative | 0 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG-Intron | INTRON A | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Age is unknown for 1 participant in each treatment group.
  Years
    number analyzed (Participants) | 62 | 62 | 124
    (all) | 48.1 (13.6) | 49.2 (12.2) | 48.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival time was defined as the time from the date of randomization to the date of disease progression or the date of death regardless of the cause. PFS was to be assessed by clinical observation, with recurrence documented by appropriate radiographic and histologic methods, and confirmed by Independent Central Review.
Time Frame: From time of randomization to time of progression or death (up to approximately 26 months)
Population: All randomized participants. Due to the early termination of this study, confirmation of PFS by Independent Central Review was not collected and; therefore, PFS could not be analyzed as planned per protocol.
Arm/Group | PEG-Intron | INTRON A
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is the time from randomization to death due to any cause. Participants were to be followed for survival every 3 months. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. After the early termination of the study, participants were followed for safety only. Although the OS analysis is not in the clinical study report due to early termination of the study, an OS ad hoc analysis was requested by the FDA and is therefore presented in this outcome measure. Below table presents the median duration of survival for participants.
Time Frame: From time of randomization to time of death (up to approximately 26 months)
Population: All treated participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PEG-Intron | INTRON A
Number analyzed (Participants) | 62 | 62
Months | NA [25.63 to NA] — NA=Median OS could not be calculated due to an insufficient number of deaths on study (i.e. median OS was not reached). NA=Upper limit OS could not be calculated due to an insufficient number of deaths on study (i.e. upper limit OS was not reached). | 23.72 [20.67 to NA] — NA=Upper limit OS could not be calculated due to an insufficient number of deaths on study (i.e. upper limit OS was not reached).
Statistical Analysis 1: Comparison: PEG-Intron vs INTRON A; Test type: Other; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.28 to 1.77] — Hazard ratio presented as PEG-Intron/INTRON A; HR <1 indicates treatment effect in favor of PEG-Intron

ADVERSE EVENTS:
Time Frame: Up to approximately 26 months
Description: Analysis population includes all participants randomized/enrolled. Adverse event preferred terms were converted from WHO-ART dictionary to the MedDRA version 10.0.
Arm/Group | PEG-Intron | INTRON A
All-Cause Mortality (participants affected / at risk) | 11/63 | 9/63
Serious Adverse Events (participants affected / at risk) | 24/63 | 19/63
Other Adverse Events (participants affected / at risk) | 61/63 | 60/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron (N=63) | INTRON A (N=63)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
TACHYARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 2 (2)
EYELID PTOSIS (Eye disorders) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
INJECTION SITE ERYTHEMA (General disorders) | 1 (1) | 0 (0)
INJECTION SITE NECROSIS (General disorders) | 2 (3) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 2 (2)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
GROIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INCISION SITE CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
WOUND ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 0 (0)
GRANULOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 2 (2) | 4 (5)
TRANSAMINASES INCREASED (Investigations) | 1 (2) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (2)
HEMIPLEGIA (Nervous system disorders) | 1 (2) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
PARAPARESIS (Nervous system disorders) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SWEAT GLAND DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ABSCESS DRAINAGE (Surgical and medical procedures) | 0 (0) | 1 (1)
ORCHIDECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron (N=63) | INTRON A (N=63)
LEUKOPENIA (Blood and lymphatic system disorders) | 7 (20) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (5) | 1 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (6) | 1 (5)
VERTIGO (Ear and labyrinth disorders) | 7 (24) | 4 (22)
EYE PAIN (Eye disorders) | 5 (13) | 5 (7)
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 (18) | 3 (4)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (9) | 7 (8)
CONSTIPATION (Gastrointestinal disorders) | 5 (10) | 9 (10)
DIARRHOEA (Gastrointestinal disorders) | 21 (65) | 15 (26)
DRY MOUTH (Gastrointestinal disorders) | 10 (36) | 15 (23)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 29 (89) | 27 (57)
VOMITING (Gastrointestinal disorders) | 20 (79) | 13 (21)
ASTHENIA (General disorders) | 22 (47) | 15 (31)
CHILLS (General disorders) | 24 (56) | 32 (76)
FATIGUE (General disorders) | 26 (186) | 28 (54)
INFLUENZA LIKE ILLNESS (General disorders) | 14 (53) | 11 (39)
INJECTION SITE ERYTHEMA (General disorders) | 10 (40) | 1 (1)
INJECTION SITE PAIN (General disorders) | 5 (6) | 1 (3)
INJECTION SITE REACTION (General disorders) | 5 (7) | 0 (0)
MALAISE (General disorders) | 6 (6) | 4 (8)
OEDEMA PERIPHERAL (General disorders) | 4 (4) | 5 (5)
PAIN (General disorders) | 11 (77) | 8 (11)
PYREXIA (General disorders) | 36 (211) | 30 (65)
BRONCHITIS (Infections and infestations) | 4 (4) | 1 (1)
INFLUENZA (Infections and infestations) | 4 (4) | 3 (4)
NASOPHARYNGITIS (Infections and infestations) | 5 (11) | 4 (6)
BODY TEMPERATURE INCREASED (Investigations) | 13 (15) | 10 (11)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 4 (4)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 4 (6)
WEIGHT DECREASED (Investigations) | 7 (9) | 5 (5)
ANOREXIA (Metabolism and nutrition disorders) | 23 (51) | 15 (20)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (7) | 7 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 (52) | 4 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 20 (81) | 15 (22)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (11)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (8) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 28 (99) | 28 (52)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14 (47) | 11 (17)
DIZZINESS (Nervous system disorders) | 17 (62) | 8 (10)
DYSGEUSIA (Nervous system disorders) | 8 (13) | 10 (10)
HEADACHE (Nervous system disorders) | 39 (231) | 33 (83)
LETHARGY (Nervous system disorders) | 8 (24) | 5 (7)
PARAESTHESIA (Nervous system disorders) | 4 (8) | 5 (5)
SOMNOLENCE (Nervous system disorders) | 2 (2) | 4 (4)
DEPRESSED MOOD (Psychiatric disorders) | 4 (5) | 1 (1)
DEPRESSION (Psychiatric disorders) | 16 (22) | 11 (16)
INSOMNIA (Psychiatric disorders) | 9 (25) | 10 (17)
SLEEP DISORDER (Psychiatric disorders) | 5 (6) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (21) | 7 (9)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (15) | 9 (16)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 14 (19) | 11 (11)
ECZEMA (Skin and subcutaneous tissue disorders) | 5 (11) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 (10) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 3 (9) | 10 (11)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (14) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 6 (10) | 3 (6)
HYPOTENSION (Vascular disorders) | 4 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed to enrollment prematurely due to sub-optimal accrual. Adverse event preferred terms were converted from WHO-ART dictionary to the MedDRA version 10.0.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator agrees not to publish or publicly present any interim results of the Protocol study without the prior written consent of the Sponsor. The Principal Investigator further agrees to provide to the Sponsor thirty (30) days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the Protocol study.